CLINICAL TRIAL: NCT04578795
Title: Effectiveness of Single Use Flexible Ureteroscopes in Treatment of Renal Stones
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Hossam Kandeel, Urology resident _ menoufia Faculty of Medicine, Menoufia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 9-2020urol
Record Dates: First submitted 2020-09-28; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Renal Stones
Keywords: Single use flexible ureteroscopy- renal stones
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pt underwent single use flexible ureteroscopy (Experimental): Patients with renal stones who will operated by single use flexible ureteroscopy
  Interventions: Device: Single use flexible ureteroscopy (PUSEN-OLIMPUS)

INTERVENTIONS:
Device: Single use flexible ureteroscopy (PUSEN-OLIMPUS) — single use flexible ureteroscopy

SUMMARY:
To study the Effectiveness of single use flexible Ureteroscopes in treatment of renal stones

DETAILED DESCRIPTION:
The miniaturization of endourological instruments and improvements in laser lithotripsy have revolutionized the approach to renal stones .

* Percutaneous nephrolithotomy (PCNL) is currently the gold standard for management of large renal calculi.
* PCNL is associated, however, with a higher complication rate, degree of risk, and longer recovery period compared with ureteroscopy - ESWL was introduced in the 1980s and quickly became the gold standard for the treatment of kidney stones . In the 1990s, URS emerged with the advantages of direct visualization and extraction of kidney calculi .
* Currently, the American Urological Association guideline recommends ESWL or URS as equivalent first-line interventions for the treatment of kidney stones < 20 mm . - The guidelines of the European Association of Urology (EAU) additionally distinguish between lower pole and non-lower pole kidney stones. They recommend both treatments as equivalent options for kidney stones of 1020 mm, but favor URS for lower pole stones if adverse factors (such as anatomy and stone composition) argue against ESWL - Flexible URS has become popular with urologists, as it is easy to learn, is associated with high stone-free rates, and is acceptable to patients .
* Firstly described in 1964 by Marshall, the uretroscope was only passively deflectable and did not include working channel. - Although the first successful procedure in humans with a ureteroscope integrating active deflection has been reported by Takayasu, it was not until 1987 that Demetrius Bagley introduced flexible ureteroscopy as we know it today ).
* we can distinguish two types of flexible URS: fiberoptic and digital flexible URS. The difference between them is the image relay and light transmission. - In fiberoptic flexible URS, light and image are transmitted in analog format through fiberoptics bundles whereas illumination in digital scopes is made by fiberoptics or by a diode (DEL) and image capture charged by a digital sensor located at the tip of the endoscope: either charged coupled device (CCD) or complementary metal oxide semiconductor (CMOS ) - In both fiberoptic and digital flexible URS, most manufacturers have models with a 3.6 Fr working channel (for irrigation and use of accessory instruments) and at least one 270° active deflection of the tip. The most recent development in flexible URS was the introduction of single use digital flexible URS .
* On the other hand the traditional reusable scopes have a fixed purchase cost, there is additional cost related to scope processing and repairs . - The cost of single-use flexible URS is defined with the initial purchase price, whereas the procedural cost of reusable flexible URS is dependent on the initial and repair cost, maintenance and scope disinfection and on the number of procedures performed before it needs to be repaired. - There is also the cost of repair and the number of procedures with a refurbished scope until it has to be replaced.

ELIGIBILITY:
Inclusion Criteria:

- All cases indicated for flexible in our department (stone kidney up to 2 cm - failed ESWL, difficult PCNL

Exclusion Criteria:

* Staghorn stones

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Clearance of renal stones | One month after operation
  the effectiveness of single use flexible ureteroscopy in treatment of renal stones in eradicate renal stones

SECONDARY OUTCOMES:
Post operative complications after flexible ureteroscopy | 3 months after operation
  Post operative complications as fever , haematuria are common after ureteroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Hossam abdelruhman kandeel, Shibīn al Kawm, Egypt